CLINICAL TRIAL: NCT05708872
Title: The Effect of Methods of Self-regulation of Mental State on Pain Perception in the Postoperative Period in Colon Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIOCHIR 01/22
Record Dates: First submitted 2022-12-27; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-12

CONDITIONS: Colonic Neoplasms; Pain, Postoperative; Hypnotherapy
Keywords: Colonic Neoplasms; Colorectal Neoplasms; Colectomy; Colorectal Surgery; Pain, Postoperative; Analgesics; Hypnosis; Autosuggestion; Mind-Body Therapies; Hypnotherapy; Psychotherapy
MeSH Terms: conditions — Colonic Neoplasms; Pain, Postoperative; Colorectal Neoplasms | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Behavioral: Autohypnosis
- Control group (Active Comparator)
  Interventions: Behavioral: Relaxing music

INTERVENTIONS:
Behavioral: Autohypnosis — Patients in the study group will receive a voice recording with hypnotic instructions with a suggestion to improve the psychophysical state.
  Arms: Study group
Behavioral: Relaxing music — Patients in the control group will receive a recording with relaxing music
  Arms: Control group

SUMMARY:
In this study, it will be investigated whether the methods of self-regulation of mental state have an effect on postoperative pain perception in colon cancer patients.

DETAILED DESCRIPTION:
According to the assumptions of psychoneuroimmunology, the improvement of mental state affects the physical improvement of patients. Numerous studies confirm the effectiveness of hypnosis and learning autohypnosis in improving the functioning of patients in terms of reducing pain and anxiety, improving the quality of sleep and mood. The study is a Prospective Randomized Controlled Trial consisting of two groups. Patients in the study group will receive a voice recording with hypnotic instructions with a suggestion to improve the psychophysical state. Patients in the control group will receive a recording with relaxing music. Depending on the randomization, patients will listen to the selected recording before being admitted to the surgical department. They will then be given a recording to listen to whenever they want. The patients will be examined four times using the Activity Change Scale, ie. before randomization, on the first day after surgery, on the 7th day after surgery and 1 month after surgery. Simultaneously the total analgesic consumption will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study
2. Age >= 18 years
3. Histopathological diagnosis of primary colon cancer without distant metastasis
4. Planned surgical treatment
5. Fluency in Polish

Exclusion Criteria:

1. Severe comorbidities with pain disorders
2. Regular use of analgesics
3. Coexistence of another neoplastic disease
4. Use of non-pharmacological pain management (including autohypnosis) prior to the study
5. Poor general condition
6. Previous colorectal surgery
7. Hearing disorders
8. No possibility of playback of the received recording

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Effect of methods of self-regulation of mental state on postoperative pain perception changes | The patient's condition will be assessed before surgery and at the following post-operative periods: the first day, the fourth day and one month after surgery.
  The timing of primary outcome measurement includes more than one time point because outcome measurements assess changes in patient status.
  The patient's condition will be assessed before surgery and at the following post-operative periods: the first day, the fourth day and one month after surgery. The measure will assess the condition over the last 24 hours on scales ranging from -10 to +10 of the Activity Change Scale.
  For pain, the score will be reviewed by asking:
  1. Which bodily sensations predominate at the site of the illness? A score of -10 indicates maximal relief; 0 neutral condition; and +10 indicates maximal pain.
  For all answers, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Effect of methods of self-regulation of mental state on mood changes | The patient's condition will be assessed before surgery and at the following post-operative periods: the first day, the fourth day and one month after surgery.
  The timing of secondary outcome measurement includes more than one time point because outcome measurements assess changes in patient status.
  The patient's condition will be assessed before surgery and at the following post-operative periods: the first day, the fourth day and one month after surgery. The measure will assess the condition over the last 24 hours on scales ranging from -10 to +10 of the Activity Change Scale.
  In terms of mood, the grade will be assessed using the following questions:
  1. What mood is prevalent? A score of -10 means a maximal increase in mood; 0 state as usual (no change); and +10 means maximal state lowered.
  For all answers, higher scores mean a worse outcome.
Effect of methods of self-regulation of mental state on anxiety changes | The patient's condition will be assessed before surgery and at the following post-operative periods: the first day, the fourth day and one month after surgery.
  The timing of secondary outcome measurement includes more than one time point because outcome measurements assess changes in patient status.
  The patient's condition will be assessed before surgery and at the following post-operative periods: the first day, the fourth day and one month after surgery. The measure will assess the condition over the last 24 hours on scales ranging from -10 to +10 of the Activity Change Scale.
  In terms of anxiety, the grade will be assessed using the following questions:
  1. What is the level of anxiety? A score of -10 means maximal calm; 0 state as usual (no change); and +10 means maximal high anxiety.
  2. How do you feel about the future? A score of -10 means maximum hope that things are going to work out; 0 status as usual (no change); and +10 means maximum anxiety about the future.
  For all answers, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Skłodowska-Curie National Research Institute of Oncology, Gliwice Branch, Gliwice, Poland

IPD SHARING:
Plan to Share IPD: No